CLINICAL TRIAL: NCT02084992
Title: A Multicenter Randomized Controlled Evaluation of Heart Failure Disease Management Using Advanced Telecommunications Within a Diverse Provider Network: The Specialized Primary and Networked Care in HF (SPAN-CHF) III Trial
Brief Title: A Study of a Technology-enabled Disease Management Program to Reduce Hospitalizations for Heart Failure
Acronym: SpanCHFIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Metro West Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Verizon2014; 11111 (Other Grant/Funding Number: Verizon Foundation)
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Congestive Heart Failure; Diastolic Heart Failure; Systolic Heart Failure
Keywords: Congestive Heart Failure; Disease management; Hospitalization
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic; Heart Failure, Systolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expanded technology disease management (Experimental): After an initial visit where the program is introduced and education regarding adherence, methods for self-monitoring and early reporting of changes in status are reviewed, patients randomized to this arm will be given tablet computers with a web-based heart failure disease management application. Patients will be asked to interact with the system daily with transmission of weight, heart rate, blood pressure and symptom reports to the nurse manager. A nurse manager will check the data daily and contact patients if any parameters exceed pre-specified parameters. Nurse managers will also touch base with the participants at regular intervals as in the control arm. In addition, educational modules will be placed onto individual tablet computers and given to each patient.
  Interventions: Other: Expanded technology disease management
- telephonic disease management (Active Comparator): After an initial visit where the program is introduced and education regarding adherence, methods for self-monitoring and early reporting of changes in status are reviewed, the nurse manager will telephone participants weekly for the first month followed by either every two weeks or monthly calls depending on clinical status with the goal of transitioning all participants to monthly calls. During these phone calls the nurse manager will focus on identifying changes in clinical condition and education reinforcement. Participants will be instructed to check and record their weight, heart rate and blood pressure daily and will be encouraged to call if there are any changes in their clinical status.
  Interventions: Other: Telephonic disease management

INTERVENTIONS:
Other: Expanded technology disease management — Tablet computers loaded with a web-based disease management program will be given to patients for the duration of the study.
  Arms: Expanded technology disease management
Other: Telephonic disease management
  Arms: telephonic disease management

SUMMARY:
This study will randomize participants with a diagnosis of congestive heart failure and at least one risk factor for hospitalization to either a tablet computer and web based disease management program or a telephone based disease management program. Both interventions are home based with heart failure education and symptom monitoring provided by nurse managers. The nurse managers are in close communication with both the participants and the participants' physicians . The components of the disease management program have been developed at Tufts Medical Center and the New England Quality Care Alliance with studies showing improved clinical outcomes, including reduced hospitalizations. The goal of this study is to transition this successful home monitoring and disease management program to a tablet computer and web-based implementation to both improve clinical outcomes (reducing hospitalizations and improving self-perceived health status) and improve provider-patient satisfaction. We hypothesize that the tablet computer based disease management will decrease heart failure hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age ≥ 18 with a primary care provider or specialist that is participating within the Collaborative Health ACO.
2. Patient able to consent
3. A diagnosis of heart failure with at least one of the following risk factors:

   * Hospitalization for heart failure within the prior year
   * NYHA class III-IV symptoms
   * Most recent BNP ≥ 300 pg/mL (or Nt-proBNP ≥ 600 pg/mL) as long as within 90 days prior to enrollment

Exclusion Criteria:

1. Acute myocardial infarction, PCI or CABG within 30 days before enrollment
2. Planned revascularization procedures, cardiac mechanical support implantation, cardiac transplantation, or other cardiac surgery within 30 days following study randomization.
3. Illness other than heart failure deemed the principal limitation to life expectancy or principal cause of disability
4. Severe angina as the principal cause of limitation
5. Uncorrected valvular disease, except where valvular regurgitation was considered to be secondary to severe left ventricular dilation, or where surgical correction is deemed excessively risky or declined by the patient.
6. Moderate to severe dementia such that unable to participate in disease management program
7. Severe visual or auditory disability such that unable to participate in disease management program
8. Hospice care
9. Listed for heart transplantation
10. No access to a working telephone
11. Homeless or no stable home environment
12. Not speaking a language in which the educational documents have been translated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2014-06; Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Number of days hospitalized for heart failure per patient-year of follow-up | 90 days

SECONDARY OUTCOMES:
All Cause Mortality | 90 days
Cardiovascular Mortality | 90 days
Number of days hospitalized for cardiovascular causes at 90 days | 90 days
Number of days hospitalized for any cause | 90 days
Change in health status as assessed by the SF-12 | 90 days
Change in self-care as assessed by the SCHFI | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Marvin A Konstam, MD, Principal Investigator — Tufts Medical Center
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - MetroWest Medical Center, Framingham, Massachusetts

REFERENCES:
- [Derived] Upshaw JN, Parker S, Gregory D, Koethe B, Vest AR, Patel AR, Kiernan MS, DeNofrio D, Davidson E, Mohanty S, Arpin P, Strauss N, Sommer C, Brandon L, Butler R, Dwaah H, Nadeau H, Cantor M, Konstam MA. The effect of tablet computer-based telemonitoring added to an established telephone disease management program on heart failure hospitalizations: The Specialized Primary and Networked Care in Heart Failure (SPAN-CHF) III Randomized Controlled Trial. Am Heart J. 2023 Jun;260:90-99. doi: 10.1016/j.ahj.2023.02.007. Epub 2023 Feb 25. PMID 36842486